CLINICAL TRIAL: NCT06060795
Title: Evaluation of the Prevalence and Evolution of Autonomic Nervous System Dysfunction for the Management of SARS-COV 2 Infection in Intensive Care Unit Patients
Brief Title: CoVID-19 Evaluation of Neurological and Autonomic Nervous System Troubles in Intensive Care Unit Patients
Acronym: COVENANT-ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D20-P014; IDRCB : 2020-A01003-36 (Other: ANSM)
Record Dates: First submitted 2020-09-23; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Symptoms; Autonomic Nervous System Dysfunction
Keywords: COVID-19; SARS-COV 2; respiratory symptoms; Autonomic Nervous system dysfunction
MeSH Terms: conditions — Signs and Symptoms, Respiratory; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Patient infected by COVID19
  Interventions: Diagnostic Test: Electro-conductance measurement
- Control group: Patient non infected by COVID19
  Interventions: Diagnostic Test: Electro-conductance measurement

INTERVENTIONS:
Diagnostic Test: Electro-conductance measurement — Interventions are done to diagnose Autonomic Nervous system Troubles
  Other Names: Tympanometry+Pupillometry

SUMMARY:
Since the spread of the COVID-19 disease, several studies have reported the presence of neurological symptoms in patients infected with SARS-CoV-2 such as dysgeusia, hypo or anosmia, hypopsia, the presence of headaches or neuralgia. It has also been described an inconsistent association, in the most severe patients, neurological disorders such as labile arterial hypertension, persistent central fever, vigilance disorders as well as a poor adaptation of the cardio vascular and respiratory systems characterized by paradoxical bradycardia and the frequent absence of polypnea in response to profound hypoxemia. These different functional signs are usually described in particular in patients with impairment of the autonomic nervous system (ANS) in connection with other neuropathological processes.

DETAILED DESCRIPTION:
Since the spread of the COVID-19 disease, several studies have reported the presence of neurological symptoms in patients infected with SARS-CoV-2 such as dysgeusia, hypo or anosmia, hypopsia, the presence of headaches or neuralgia. It has also been described an inconsistent association, in the most severe patients, neurological disorders such as labile arterial hypertension, persistent central fever, vigilance disorders as well as a poor adaptation of the cardio vascular and respiratory systems characterized by paradoxical bradycardia and the frequent absence of polypnea in response to profound hypoxemia. These different functional signs are usually described in particular in patients with impairment of the autonomic nervous system (ANS) in connection with other neuropathological processes.

Currently, there are few studies interesting by the neurological complications of patients with SARS-CoV-2, the mechanisms involved in its migration to target sites and the processes leading to damage by direct injury or related to neuro-inflammatory processes of the CNS and in particular of the brainstem, responsible for the regulation of the ANS.

The main objective of the study conducted is therefore to evaluate the prevalence and the evolution of autonomic nervous system dysfunction and its impact in patients with SARS-CoV-2 infection hospitalized in intensive care Unit (ICU) confirmed by the obtaining a positive RT-PCR (2nd PCR carried out 3 days after the first in the event of a negative first result). This dysfunction of Autonomic Nervous System will be diagnosed on the basis of a multimodal assessment including spectral analysis of heart rate variability, the tone, pupillary reactivity and tympanometry, the measurement of skin electro-conductance, evaluation of diaphragmatic function and analysis of electro-encephalographic characteristics.

This population of patients will be compared with a control group of subjects admitted in ICU for the management of a suspected SARS-CoV-2 infection with a diagnosis excluded on the basis of a set of clinical and biological and ultrasound arguments associated with two RT-PCRs on negative respiratory samples taken 3 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, hospitalized in an intensive care unit for the management of a suspected SARS-CoV-2 infection diagnosed by reference examination (PCR on nasopharyngeal Sample)
* Patient affiliated or benefiting from a social security system,
* Consent obtained from the trusted person, or close person or parent, under the conditions provided by the article L.1122-1-1 of the "CSP"
* Patient who has given consent to participate.

Exclusion Criteria:

* Bad command of French language or state incompatible with the patient's understanding and / or enlightened adherence to the study protocol
* Adults who are the subject of legal protection or unable to express their consent
* Minors
* Lack of possible collection of signed informed consent
* History of progressive and / or degenerative neurological pathology
* Pregnant women, parturients and nursing mothers
* Therapeutic limitation decision made before inclusion of patient
* Persons deprived of their liberty by a court or administrative decision, persons undergoing psychiatric care (article L1121-6)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The 'experimental group' population in question consisted of patients over 18 years of age at the time of inclusion, admitted to an intensive care unit or intensive care unit for the management of an established SARS-CoV-2 infection.
  The 'control group' population consisted of adult patients, male or female, admitted to an intensive care unit or intensive care unit for the management of respiratory symptoms requiring continuous monitoring but whose final diagnosis was based on several clinical-biological and radiological a posteriori, is not related to SARS-CoV-2 infection and has two negative RT-PCRs for SARS-CoV-2 performed three days apart (1st PCR performed on admission to the ward and re-sampling in case of first negative PCR).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Prevalence and ANS dysfunction defined by the presence of the following criteria, isolated or associated | Day1, Day3, Day7, Day14, Day21
  * Criterion 1: A significant change in the LF / HF ratio and AUCHR compared to baseline and control group
  * Criterion 2: A significant change in the measurement of average skin conductances on the hands and feet in COVID-19 patients compared to baseline and control group
  * Criterion 3: A significant change in basic tone and pupillary reactivity to light stimuli and pain in COVID-19 patients compared to baseline measures and control group
  * Criterion 4: A significant change in the tympanic reflex observed in COVID-19 patients compared to baseline and control group,
  * Criterion 5: Presence of significant changes in EEG pattern and evolution between COVID-19 patients and control group

SECONDARY OUTCOMES:
Presence of an ARDS defined by the new definition of "Berlin" of acute respiratory distress syndrome (ARDS), | Day1, Day3, Day7, Day14, Day21
  proposed distinguished according to the PaO2 / FiO2 ratio measured in the presence of a positive external expiratory pressure (PEPe) of at least 5 cmH2O, three levels of ARDS severity in minimal (200 <PaO2 / FiO2 ≤ 300 mmHg), moderate (100 <PaO2 / FiO2 ≤ 200 mmHg) and severe (PaO2 / FiO2 ≤ 100 mmHg),
Mortality at 1 month | Month 1
  - Vital status at 30 days
Mortality at 6 months | Month 6
  - Vital status at 6 months
Sequential Organ Failure Assessment (SOFA score) | Day1, Day3, Day7, Day14, Day21
  SOFA score: grade the organ function or failure rate, from 0 to 24, severity increases as the score increases.
Total duration of mechanical ventilation, ventilatory weaning, curarization, | Day 21
  Total time of mechanical ventilation, weaning and use of neuromuscular blockade

CONTACTS AND LOCATIONS:
Overall Officials: DANIEL Matthieu, MD, PhD, Principal Investigator — Centre hospitalier Sainte Anne
Locations (1):
- Centre Hospitalier Sainte-Anne, Paris, France

IPD SHARING:
Plan to Share IPD: No